CLINICAL TRIAL: NCT07072858
Title: Prognostic Value of Cardiac Magnetic Resonance Parameters in Patients With ST-Segment Elevation Myocardial Infarction
Brief Title: Using Cardiac MRI to Predict Outcomes in Patients With STEMI
Acronym: CMR-RISK-STEMI
Status: Recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, XIN A, Dr, Chinese PLA General Hospital
Other Study IDs: S2025-061-01
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-01

CONDITIONS: Myocardial Infarction (MI); ST Segment Elevation Myocardial Infarction (STEMI); Magnetic Resonance Imaging (MRI); Heart Ventricles; Artificial Intelligence (AI); Prognosis; Ventricular Dysfunction
Keywords: ST Segment Elevation Myocardial Infarction; Cardiac Magnetic Resonance Imaging; Cardiac Strain Imaging; Machine Learning; Image Analysis; Survival Analysis; Multimodal Imaging
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction; Ventricular Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- STEMI Patients Undergoing CMR After PCI
  Interventions: Diagnostic Test: Cardiac Magnetic Resonance Imaging (CMR)

INTERVENTIONS:
Diagnostic Test: Cardiac Magnetic Resonance Imaging (CMR) — Cine CMR imaging was performed with steady-state free precession covering short axis continuously from the mitral annulus to the apical level in the 2-, 3- and 4- chamber views using the following parameters: repetition time (TR) = 3.73 ms, echo time (TE) = 1.87 ms, flip angle = 60°, slice thickness 8.0 mm. Cine images of all included patients were acquired prior to contrast administrations. Late gadolinium enhancement images (LGE) images were obtained 10-15 minutes after intravenous injection of gadolinium (0.1 mmol/kg at 3ml/s) at end-diastolic phase on the short axis (TR=6.09 ms; TE= 3.0 ms; flip angle 60°; thickness 8.0 mm) with breath-hold phase-sensitive segmented inversion recovery (PSIR) fast field echo sequence. T2-weighted sequence was performed using turbo spin-echo (TSE)-sequence (TR=1714-2000 ms; TE=8.04 ms; slice thickness 8.0 mm) to estimate myocardial edema. Images were analyzed on freely available validated cardiovascular image analysis software CVI42 (Circle Cardiovas

SUMMARY:
This prospective, multicenter observational study aims to evaluate the prognostic value of a comprehensive set of cardiac magnetic resonance (CMR) imaging parameters in patients with ST-segment elevation myocardial infarction (STEMI) undergoing primary percutaneous coronary intervention (PCI). The study integrates advanced artificial intelligence (AI) techniques to extract and analyze high-dimensional imaging features from multiple CMR sequences-including cine, strain mapping, and functional sequences-going beyond traditional measures such as infarct size or microvascular obstruction.

The primary objective is to identify novel prognostic markers from routinely acquired CMR images that reflect myocardial structure, function, and mechanical deformation (strain), and to assess their association with long-term clinical outcomes. In addition to standard parameters, the study includes a detailed evaluation of left and right ventricular systolic and diastolic volumes, ejection fractions, and biventricular strain components (including longitudinal, circumferential, and radial strain), as well as left and right atrial volumes, emptying fractions, and reservoir/conduit/booster strain indices.

Approximately 1000 STEMI patients will undergo CMR scanning within one week after PCI. The imaging data will be subjected to AI-based feature extraction and dimensionality reduction algorithms to uncover latent patterns associated with adverse outcomes. Patients will be followed for up to three years for the occurrence of major adverse cardiovascular events (MACE), including cardiovascular death, recurrent myocardial infarction, and heart failure hospitalization.

The central hypothesis is that comprehensive CMR functional and strain-derived parameters, when analyzed using AI-driven models, offer independent and incremental prognostic value beyond conventional clinical risk factors. This study seeks to establish a data-driven, multimodal imaging framework for personalized risk stratification in STEMI patients, potentially enabling more precise post-infarction management strategies.

No investigational treatment is involved. All imaging and clinical data are collected as part of routine care and analyzed retrospectively for outcome prediction.

DETAILED DESCRIPTION:
This is a prospective, multicenter observational study designed to investigate the prognostic value of comprehensive cardiac magnetic resonance (CMR) imaging parameters in patients with ST-segment elevation myocardial infarction (STEMI) who undergo primary percutaneous coronary intervention (PCI). The study focuses on leveraging artificial intelligence (AI)-based analysis to extract predictive features from a wide range of standard and advanced CMR sequences, aiming to identify imaging-derived biomarkers that provide independent and incremental value in forecasting long-term cardiovascular outcomes.

Traditional CMR indicators such as infarct size, left ventricular ejection fraction (LVEF), and microvascular obstruction (MVO) have demonstrated utility in post-MI risk stratification. However, these parameters do not fully exploit the wealth of information embedded within the full CMR dataset, especially data reflecting myocardial and atrial mechanics. In this study, we apply advanced computational methods-including radiomics, machine learning, and survival modeling techniques-to analyze multidimensional features extracted from routine, non-contrast CMR sequences.

CMR image acquisition includes short-axis cine imaging and dedicated functional sequences allowing for the quantification of bi-ventricular and bi-atrial function and deformation. Specifically, the following parameters are collected and analyzed:

* Left Ventricular (LV) Parameters LV End-Diastolic Volume (LVEDV) LV End-Systolic Volume (LVESV) LV Stroke Volume (LVSV) LVEF Global Longitudinal Strain (LVGLS) Global Circumferential Strain (LVGCS) Global Radial Strain (LVGRS)
* Right Ventricular (RV) Parameters RVEDV RVESV RVSV RV Mass RVEF RVGLS, RVGCS, RVGRS
* Left Atrial (LA) Parameters Maximum Volume (LAVmax) Pre-Atrial Contraction Volume (LAVpac) Minimum Volume (LAVmini) Total, Passive, and Booster Emptying Fractions (LAEF) Reservoir, Conduit, and Booster Strain
* Right Atrial (RA) Parameters RAVmax RAVpac RAVmini Total, Passive, and Booster RAEF RA Reservoir, Conduit, and Booster Strain All images are analyzed by trained imaging specialists using semi-automated tools (e.g., CVI42) for myocardial and atrial contouring. The left ventricular myocardium is segmented at the end-diastolic phase, and regions of interest (ROIs) are exported for radiomic analysis using ITK-SNAP and PyRadiomics. Preprocessing includes voxel size resampling, normalization, and gray-level discretization.

To ensure reliability and minimize redundancy, feature selection is performed in several stages. First, features with intra- and inter-observer intraclass correlation coefficients (ICC) ≥ 0.75 are retained. Second, highly collinear features are removed using correlation thresholding. Third, feature importance is assessed via random survival forests (RSF), followed by least absolute shrinkage and selection operator (LASSO) Cox regression to construct an optimized feature set. Selected features are used to calculate a radiomics-based risk score (RAD score), which is incorporated into survival models.

Patients are divided into a training and validation cohort using stratified random sampling based on MACE incidence. The primary outcome is the occurrence of major adverse cardiovascular events (MACE), including cardiovascular death, reinfarction, and heart failure hospitalization. Prognostic models are developed using multivariable Cox regression and evaluated using Harrell's concordance index (C-index), calibration plots, and time-dependent receiver operating characteristic (ROC) curves. Risk stratification analyses are conducted across subgroups defined by conventional imaging markers (e.g., infarct size, LVEF, MVO).

The analysis pipeline is implemented using R software, and internal validation is performed to assess model stability. Multiple imputation is used to address missing data, and sensitivity analyses are conducted to test the robustness of the predictive models under various assumptions. No experimental intervention or investigational drug is administered in this study; data collection is non-interventional and integrated into routine clinical care.

The anticipated contribution of this study is to establish a multimodal, AI-enhanced imaging framework that enables individualized post-STEMI risk assessment using routinely available CMR data. By going beyond visually assessed or conventional parameters, this study may uncover novel patterns of myocardial and atrial dysfunction predictive of long-term outcomes. Furthermore, the use of non-contrast imaging sequences enhances the generalizability and safety of the proposed risk evaluation method.

The protocol is approved by the institutional ethics committee. Quality control includes standardized image acquisition and analysis procedures across centers. Data processing follows pre-specified standard operating procedures (SOPs) for image segmentation, radiomic feature extraction, and modeling. Manual and automated data checks are implemented to ensure consistency and accuracy. The imaging core lab and analytic team remain blinded to outcome data during feature extraction and model construction phases.

By combining cutting-edge image analysis with real-world clinical data, this study aims to inform future CMR-based guidelines for post-infarction care and to facilitate clinical translation of advanced imaging biomarkers into personalized cardiology.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years

Diagnosed with ST-segment elevation myocardial infarction (STEMI), defined as chest pain with ST-segment elevation on ECG and elevated cardiac troponin levels

Underwent primary percutaneous coronary intervention (PCI)

Able to undergo cardiac magnetic resonance (CMR) imaging within 7 days post-PCI

Provided written informed consent

Exclusion Criteria:

* Contraindications to CMR (e.g., severe claustrophobia, implanted cardiac defibrillators or non-compatible pacemakers)

History of revascularization therapy (PCI or CABG) within the previous 6 months

Severe valvular heart disease or known cardiomyopathy

Presence of bundle branch block or fascicular block that interferes with image interpretation

Known allergy to gadolinium-based contrast agents (for those undergoing contrast-enhanced sequences)

Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m² (if contrast use is anticipated)

Pregnant or breastfeeding women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients diagnosed with ST-segment elevation myocardial infarction (STEMI) who are treated with primary percutaneous coronary intervention (PCI). Eligible participants must be able to undergo cardiac magnetic resonance (CMR) imaging within one week of PCI. Patients are recruited from cardiology departments at high-volume centers with established CMR capabilities. The population includes both men and women, aged 18 to 80 years, representing a typical real-world cohort of STEMI patients in clinical practice. Patients with significant comorbidities, contraindications to MRI, or recent prior revascularization are excluded to ensure reliable image interpretation and outcome attribution.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Major Adverse Cardiovascular Events (MACE) | From the date of CMR imaging to the first occurrence of MACE during follow-up (maximum of 5 years)
  Major Adverse Cardiovascular Events (MACE) is defined as a composite outcome including cardiovascular death, non-fatal myocardial infarction, and hospitalization for heart failure. The occurrence of MACE during follow-up will be used to assess the prognostic value of CMR-derived parameters and AI-based imaging features.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided